CLINICAL TRIAL: NCT06981013
Title: Effects of Balance-based Torso Weighting on Muscle Activation During Balance Tests in Individuals With and Without Multiple Sclerosis
Brief Title: Effects of Torso Weighting on Muscle Activation During Balance Tests in Individuals With and Without Multiple Sclerosis
Acronym: BBTW-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of St. Augustine for Health Sciences (Other)
Responsible Party: Principal Investigator, Evan M. Pucillo, PT, DPT, EdD, Director of Research, University of St. Augustine for Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-1101-275
Record Dates: First submitted 2025-04-25; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; muscle activation; ankle muscles; balance vest
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: 20 participants with multiple sclerosis and 20 participants without multiple sclerosis in a Quasi experimental design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple Sclerosis Arm (Experimental): Without and with balance-based torso weighting
  Interventions: Other: balance based torso weighting
- Healthy Control Arm (Active Comparator): Without and with balance-based torso weighting
  Interventions: Other: balance based torso weighting

INTERVENTIONS:
Other: balance based torso weighting — The intervention in this study is the Balance-Based-Torso-Weighting (BBTW) which will be applied on individuals with MS and healthy controls. It involves the strategic placement of weights based on the assessment of the loss of balance in three dimensions: anterior-posterior, lateral, rotational to counteract the balance loss.4 The BBTW Evaluation Tool Kit will be used to determine the location of the weights. It consists of an adjustable testing vest; rigid orthotic; five pounds worth of weights divided into 1/16, 1/8, 1/4, 1/2 lb. increments; and exam evaluation forms (www.motiontherapeutics.com).

SUMMARY:
Rationale: The Balance-Based Torso-Weighting (BBTW) is a patented evaluation system that uses strategic placement of small or lightweight weights on the trunk to improve balance and stability. BBTW has been found to improve the upright mobility of people with multiple sclerosis, however the mechanism underlying the improvement of balance and gait is still unknown.1-2 Purpose: The purpose of this study is to investigate the immediate effects of BBTW on muscle activation of tibialis anterior and gastrocsoleus and sway using electromyography and force plates during balance tests in people with MS and healthy controls?

DETAILED DESCRIPTION:
Research Questions:

Question #1 - Is there a difference in EMG within postural muscles (tibialis anterior and gastrocsoleus) and between healthy and MS when not wearing weighted vest with eyes open? Question #2 - Is there a difference in EMG within postural muscles (tibialis anterior and gastrocsoleus) and between healthy and MS when not wearing weighted vest with eyes closed? Question #3 - Is there a difference in EMG within postural muscles (tibialis anterior and gastrocsoleus) and between healthy and MS when wearing weighted vest eyes open? Question #4 - Is there a difference in EMG within postural muscles (tibialis anterior and gastrocsoleus) and between healthy and MS when wearing weighted vest eyes closed? Question #5 - Is there a difference in SWAY within postural muscles (tibialis anterior and gastrocsoleus) and between healthy and MS when not wearing weighted vest with eyes open? Question #6 - Is there a difference in SWAY within postural muscles (tibialis anterior and gastrocsoleus) and between healthy and MS when not wearing weighted vest with eyes closed? Question #7 - Is there a difference in SWAY within postural muscles (tibialis anterior and gastrocsoleus) and between healthy and MS when wearing weighted vest eyes open? Question #8 - Is there a difference in SWAY within postural muscles (tibialis anterior and gastrocsoleus) and between healthy and MS when wearing weighted vest eyes closed? Research Design: Quasi-experimental design

ELIGIBILITY:
Inclusion Criteria for Individuals with Multiple Sclerosis group:

* self-reported diagnosis of multiple sclerosis (MS)
* age 18 to 75 years old
* able to communicate in English
* able to provide informed consent
* able to tolerate up to three hours of testing with rest breaks
* able to walk 20 meters with or without assistive device and without resting (equivalent to Expanded Disability Status Scale of 6.5 or less).

Inclusion criteria for the Healthy Control group:

* able to communicate in English
* able to provide informed consent
* physical criteria that matched each participant with MS which included age (within 7 years), height (within 12.7 cm [5 in]), mass (within 9.1 kg [20 lb]) and sex.

Exclusion Criteria for Individuals with Multiple Sclerosis group:

* exacerbation of MS within the past two months
* had a diagnosis of a concurrent neurological disorder (head injury, stroke, Parkinson's disease, etc.)
* reported pain that could be exacerbated by external perturbations during standing.

Exclusion Criteria for Healthy control group:

* Known diagnoses
* current pain that could affect balance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Muscle Activation of B lateral gastrocnemius and tibialis anterior | Baseline and study completion, after an average of three hours
  Noraxon EMG will be used to measure muscle activation
Postural Sway as measured by center of pressure displacement | Baseline and study completion, after an average of three hours
  Kistler Force Plate will be used center of pressure displacement in the x and y axis

CONTACTS AND LOCATIONS:
Overall Officials: Amie Marie F Jasper, DPT, PhD, Principal Investigator — USAHS
Locations (1):
- University of St. Augustine for Health Sciences, Saint Augustine, Florida, United States